CLINICAL TRIAL: NCT04932902
Title: ManAgement of pRiapiSm and Its Impact on Outcomes: an International Register
Brief Title: ManAgement of pRiapiSm and Its Impact on Outcomes
Acronym: MARS
Status: Enrolling by invitation | Type: Observational
Sponsor: Policlinic Hospital "G. Rodolico" (Other)
Collaborators: European Association of Urology Research Foundation (Other)
Responsible Party: Principal Investigator, Giorgio Ivan Russo, Prof. Giorgio Ivan Russo, Policlinic Hospital "G. Rodolico"
Other Study IDs: 122/2021
Record Dates: First submitted 2021-06-13; First posted 2021-06-21 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Priapism
MeSH Terms: conditions — Priapism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Priapism is a urological emergency that is defined as a prolonged penile erection lasting more than 4 h, remaining despite orgasm and in the absence of sexual stimulation. There are three sub-types of priapism: Ischaemic, non- ischaemic and stuttering. The most common (95% cases) of these is ischaemic priapism (IP), which represents a compartment syndrome of the corpus cavernosa with minimal or no arterial flow into the penis. It causes time-dependent smooth muscle damage that can result in significant morbidity (including, permanent erectile dysfunction (ED), penile shortening, penile curvature and loss of girth) with- out prompt intervention.

Unlike ischemic priapism, non-ischemic priapism is not a urologic emergency, both the American Urological Association (AUA) and the European Association of Urology (EAU) recommend conservative, non-operative, management for the treatment of NIP. Spontaneous resolution has been documented to occur in 62% of patients [1].

Despite the very high burden of priapism and its time-dependent adverse effect on erectile function, few studies have comprehensively defined the clinical epidemiology of this complication nor have any compared sexual dysfunction in men with SCD with that in those without it. Evidence-based treatment strategies for priapism are currently lacking, especially in terms of sexual function.

However, despite the various publications in the literature, even today the published studies show considerable bias, in terms of sample size, evaluation of reproducible outcomes, use of internationally validated questionnaires, well-defined follow-up evaluation, as well as the evaluation of outcome after medical or surgical treatment. For this reason, the purpose of this international register is precisely to shed light on what may be the responses to medical surgical treatment in patients with priapism, but in particular to set up a rational data collection that has solid scientific bases.

DETAILED DESCRIPTION:
Aims and objectives

Based on the previous premises, the aim of our study is to evaluate the impact of the management of priapism from a sexual and clinical long-term outcomes point of view.

Sexual outcomes will be assessed by measured questionnaire (e.g. IIEF-15) at 3-6 months after priapism.

Clinical outcomes will be registered as rates of resolution of acute priapism within 30' after the onset of treatment (defined as no need for further non-surgical/surgical interventions to resolve priapism episode), corporal injury (fibrosis or necrosis), adverse events including erectile dysfunction, penile curvature/Peyronie's disease, requirement for surgical management of priapism.

Sample size calculation

Since the study is designed as a prospective data collection through a registry, and since there are no comparative analyses between different groups, it is not possible to identify a priori sample size. However, considering that the largest case history on the field of priapism amounts to a total of 112 patients [3], we believe that collecting data from a total of 200 patients is sufficient in order to obtain scientifically reliable results with a high scientific profile.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Priapism

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with priapism: ischemic, non-ischemic or stuttered.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
IIEF-5 at 3 months | 3 months
  Sexual function as reported by patient or measured by questionnaire

SECONDARY OUTCOMES:
IIEF-5 at 6 months | 6 months
  Sexual function as reported by patient or measured by questionnaire
Requirement for surgical management of priapism | Within 1 month
  Requirement for surgical management of priapism
Adverse events including erectile dysfunction, penile curvature/Peyronie's disease | 6 months
  Adverse events
Resolution | 30 minutes
  Resolution of acute priapism within 30' after the onset of treatment (defined as no need for further non-surgical/surgical interventions to resolve priapism episode)

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Ivan Russo, MD, Principal Investigator — Associate Professor, Urology Unit, Policlinic Hospital G. Rodolico
Locations (5):
- Italy (4):
  - Giorgio Ivan Russo, Catania, CT
  - University of Florence, Florence
  - University of Torino, Torino
  - University of Varese, Varese
- Serviço de Urologia, Centro Hospitalar Universitário São João, Porto, Portugal, Porto, Portugal